CLINICAL TRIAL: NCT05995509
Title: The Effect of Number of Micro-osteo-perforations on the Rate of Tooth Movement: A Randomized Controlled Trial.
Brief Title: The Effect of Number of Micro-osteo-perforations on the Rate of Tooth Movement.
Acronym: MOPs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehman Medical Institute - RMI (Other)
Collaborators: Gandhara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPSP/REU/DSG-2017-026-2176
Record Dates: First submitted 2023-05-13; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Orthodontic Tooth Movement
Keywords: Micro-osteo-perforations; orthodontic tooth movement; clinical trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 MOPs group (Active Comparator): The subjects under a split mouth intervention on the experimental side will undergo 3 micro-osteo-perforations (creating small holes in the buccal cortical bone) to assess the rate of tooth movement.
  Interventions: Procedure: Micro-osteo-perforations
- 1 MOP group (Experimental): the subjects under the split mouth intervention on the control side will undergo 1 micro-osteo-perforation in comparison to the experimental side.
  Interventions: Procedure: Micro-osteo-perforations

INTERVENTIONS:
Procedure: Micro-osteo-perforations — small perforations drilled in Alveolar bone, adjacent to site of tooth movement.

SUMMARY:
The objective of this split mouth trial is to compare mean canine retraction with one Micro-osteo-perforation (MOP) against three MOPs among Class II division I orthodontic patients after one month of intervention.

DETAILED DESCRIPTION:
One of the main concerns for orthodontists and patients who seek orthodontic therapy is the prolonged treatment time. A commitment of about 18-24 months makes decision making difficult for many patients. The prolonged treatment time is also a potential factor leading to complications like white spot lesions, root resorption, gingivitis and periodontitis. Different techniques to speed up tooth movement have been used in orthodontics. Micro-osteo-perforations is one of the new ways to expedite tooth movement. Previous trials of MOP (Micro-osteo-perforations) to expedite tooth movement had certain shortcomings including the lack of details of randomization. Further studies with variation in the number and frequency of MOPs over a longer duration were recommended. It also raises a curiosity if reducing the number of MOPs would be equally effective in accelerating the canine retraction. Hence, the purpose of this split mouth trial was to investigate the effect of number of MOPs on the rate of canine retraction.

The objective of this split mouth trial is to compare mean canine retraction with one MOP against three MOPs among Class II division I orthodontic patients after one month of intervention.

STUDY DESIGN: Split-mouth parallel arm randomized control trial.

ELIGIBILITY:
Inclusion Criteria: All male and female patients in an age range of 12-25 years requiring bilateral first premolar extraction in maxillary arch.

-

Exclusion Criteria:

1. Patients with any sort of systemic disease.
2. Radiographic evidence of bone loss.
3. History of periodontal therapy
4. Active periodontal disease.
5. Patients with a history of smoking of five years or more.
6. Patients with active gingivitis and Caries.
7. Attrition of canine cusp.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The rate of tooth movement (canine retraction) | The movement of canines on both sides will be measured after 30 days of 150g of force application on the intervention and control side.
  The canine retraction will be measured from a mid-palatine line drawn on the pre treatment and post MOP dental cast. Further perpendicular lines will be drawn towards the distal surface of canine and the mesial surface of the second premolar. The Canine retraction will be measured as the difference between the two lines measured in millimetres. The clinical significance will be set at 50% or more of the rate of canine retraction of the control side.

SECONDARY OUTCOMES:
Pain associated with MOPs | In the surgery after the procedure is completed and just before the patient was sent home.
  The pain or discomfort to the patient will be assessed using a Baker's visual analogue scale on the control and the experimental sides. The scale will be calibrated in millimetres from 0-10 with 0 denoting no pain and 10 denoting worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Tajik, FCPS, Study Chair — Sardar Begum Dental College
Locations (1):
- RMI, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No